CLINICAL TRIAL: NCT06168409
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Effect of Baxdrostat on Ambulatory Blood Pressure in Participants With Resistant Hypertension
Brief Title: A Study to Investigate the Effect of Baxdrostat on Ambulatory Blood Pressure in Participants With Resistant Hypertension
Acronym: Bax24
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6970C00009; 2023-507640-36-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Resistant Hypertension
Keywords: Hypertension; Resistant hypertension; Blood pressure; Baxdrostat; CIN-107; Aldosterone; Aldosterone synthase; Aldosterone synthase inhibitor
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 mg baxdrostat (Experimental): 2 mg baxdrostat administered orally, once daily (QD).
  Interventions: Drug: Baxdrostat
- Placebo (Placebo Comparator): Placebo administered orally, once daily (QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat tablet administered orally, once daily (QD). Unit dose strength:
  • 2 mg per tablet.
  Other Names: CIN-107
  Arms: 2 mg baxdrostat
Drug: Placebo — Placebo tablet matching baxdrostat, administered orally, once daily (QD).
  Arms: Placebo

SUMMARY:
This is a Phase III, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety, tolerability and the effect of 2 mg Baxdrostat vs. placebo, administered QD orally, on the reduction of SBP, measured by average 24-hour ABPM in 212 participants with rHTN (defined as seated SBP ≥ 140 mmHg at Screening and mean ambulatory SBP ≥ 130 mmHg at baseline, despite a stable regimen of ≥ 3 antihypertensive agents, one of which is a diuretic).

DETAILED DESCRIPTION:
This is a Phase III, multicentre, randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety, tolerability and the effect of 2 mg baxdrostat versus placebo, administered once a day (QD) orally, on the reduction of ambulatory SBP in participants with rHTN, defined as BP targets not being achieved in an individual despite the use of at least 3 antihypertensive agents of different classes (at maximum tolerated dose in the judgement of the Investigator), one of which is a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years old, at the time of signing the informed consent.
* Mean seated SBP on AOBPM of ≥ 140 mmHg and < 170 mmHg at Screening.
* Have a stable regimen of ≥ 3 antihypertensive medications, from different therapeutic classes (at least one must be a diuretic), at maximum tolerated dose in the judgement of the Investigator, for at least 4 weeks prior to screening. Beta blockers used to treat other conditions (ie, migraine, HF, coronary artery disease) should not be counted as an antihypertensive medication for the purpose of qualifying for this study.
* Have eGFR ≥ 45 mL/min/1.73 m2 at Screening.
* Serum potassium (K+) level ≥ 3.5 and < 5.0 mmol/L at Screening, determined as per central laboratory
* Randomization Criteria: mean ambulatory SBP of ≥ 130 mmHg at randomisation.

Exclusion Criteria:

* Mean seated SBP on AOBPM ≥ 170 mmHg.
* Mean seated DBP on AOBPM ≥ 110 mmHg.
* Serum sodium level < 135 mmol/L at Screening, as per central laboratory.
* Participant has the following known secondary causes of hypertension: renal artery stenosis, uncontrolled or untreated hyperthyroidism, uncontrolled or untreated hypothyroidism, pheochromocytoma, Cushing's syndrome, aortic coarctation.
* New York Heart Association functional HF class IV.
* Persistent atrial fibrillation.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ambulatory 24-hour average SBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory 24-hour average SBP at Week 12.

SECONDARY OUTCOMES:
Change from baseline in ambulatory night-time average SBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory night-time average SBP at Week 12.
Change from baseline in ambulatory daytime average SBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory daytime average SBP at Week 12.
Change from baseline in seated SBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on seated SBP at Week 12.
Participants achieving ambulatory 24-hour average SBP of < 130 mmHg | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on achieving ambulatory 24-hour average SBP < 130 mmHg at Week 12.
Change from baseline in ambulatory 24-hour average DBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory 24-hour average DBP at Week 12.
Change from baseline in ambulatory night-time average DBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory night-time average DBP at Week 12.
Change from baseline in the average ambulatory daytime average DBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on ambulatory daytime average DBP at Week 12.
Change from baseline on seated DBP | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo on seated DBP at Week 12.
Participants achieving a nocturnal SBP dipping of ≥ 10% | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg versus placebo in the nocturnal dipping pattern at Week 12.

CONTACTS AND LOCATIONS:
Locations (92):
- United States (16):
  - Research Site, Surprise, Arizona
  - Research Site, Hollywood, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, The Bronx, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Brownsville, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Lampasas, Texas
- Argentina (7):
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Córdoba
  - Research Site, Lanús Este
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, San Vicente
- Australia (2):
  - Research Site, Clayton
  - Research Site, Perth
- Research Site, Ghent, Belgium
- Research Site, Sofia, Bulgaria
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, North Vancouver, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Terrebonne, Quebec
- Czechia (4):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Broumov
  - Research Site, Louny
- Germany (4):
  - Research Site, Bad Homburg
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Kaiserslautern
- Greece (3):
  - Research Site, Athens
  - Research Site, Attica
  - Research Site, Thessaloniki
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Kalocsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
- Malaysia (3):
  - Research Site, Kota Bharu
  - Research Site, Muar town
  - Research Site, Sarawak Miri
- Philippines (2):
  - Research Site, Angeles City
  - Research Site, Iloilo City
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Research Site, Riyadh, Saudi Arabia
- Slovakia (3):
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Svidník
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Durban
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santa Coloma de Gramenet
  - Research Site, Terrassa (Barcelona)
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, New Taipei City
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Odunpazari
- United Kingdom (7):
  - Research Site, Corby
  - Research Site, London
  - Research Site, Prescot
  - Research Site, Swindon
  - Research Site, Thetford
  - Research Site, Weston-super-Mare
  - Research Site, Yate
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Dwyer JP, Maklad N, Vedin O, Monyak J, Myte R, Chertow GM, Heerspink HJL, Little DJ. Efficacy and Safety of Baxdrostat in Participants with CKD and Uncontrolled Hypertension: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Sep 6. doi: 10.1681/ASN.0000000849. Online ahead of print. No abstract available. PMID 40913594